CLINICAL TRIAL: NCT07180576
Title: The FORCE Trial Pilot
Brief Title: The FORCE Trial Pilot: Fish Oil-enriched Nutrition for Radiotherapy in Cancer of the hEad and Neck
Acronym: FORCE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anna Arthur, PhD (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor-Investigator, Anna Arthur, PhD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00161711; UKHSRR number: 4907 (Other: University of Kansas Medical Center)
Record Dates: First submitted 2025-09-05; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Head &Amp;Amp; Neck Squamous Cell Carcinoma
Keywords: nutrition; head and neck cancer; nutrition supplement; nutrition trial; fish oil; cancer patient; sarcopenia; nutrition impact symptoms; body composition; cancer; oncology; fatty acid; cancer survivor; oral nutrition supplement; supportive care
MeSH Terms: conditions — Head and Neck Neoplasms; Sarcopenia; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supplemental drink (Experimental): This is a single-arm design; comparisons are pre- vs. post-intervention or against feasibility thres
  Interventions: Behavioral: Nutrition counseling; Drug: Fresubin Supportan

INTERVENTIONS:
Behavioral: Nutrition counseling — Weekly standardized nutrition counseling will be provided by a study RDN to promote adherence and address barriers to adherence, acceptability, and adverse events. The RDN will also document any changes to the CRT regimen and hospitalizations.
Drug: Fresubin Supportan — Two bottles per day of Fresubin Supportan, a fish oil-enriched high calorie, high protein oral nutrition supplement.

SUMMARY:
en-label, proof-of-concept study designed to evaluate the feasibility, safety, and acceptability of a prophylactic fish oil-enriched nutritional supplement (Fresubin Supportan) in patients with head and neck cancer (HNC) undergoing curative-intent chemoradiotherapy (CRT) at the University of Kansas Medical Center. The study involves daily supplementation starting two weeks prior to CRT and continuing throughout CRT, alongside weekly nutrition counseling.

DETAILED DESCRIPTION:
This will be a single-arm, open-label, proof-of-concept (PoC) study conducted at the University of Kansas Medical Center (KUMC). The overarching goal is to assess feasibility, safety, acceptability, and preliminary efficacy signals of pre- and peri-CRT fish oil-enriched drink (Fresubin Supportan) in 15 HNC patients undergoing definitive CRT. The intervention duration will be ~8.5-9 weeks (2 weeks pre-RT + ~6.5-7 weeks during CRT). The intervention includes weekly nutrition counseling from a Registered Dietitian Nutritionist (RDN) and biospecimen collection for fatty acid analysis, FADS1/2 genotyping, and long-term banking for future biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with Stage I - IV oral cavity, hypopharyngeal, oropharyngeal, or laryngeal cancer
* Age 18+
* Planned for definitive radiotherapy with or without surgery and chemotherapy

Exclusion Criteria:

* Metastatic disease
* Prior head/neck RT
* Presence of malnutrition at diagnosis per ASPEN criteria
* Prior cancer within 3 years (except non-melanoma skin cancer and cervical carcinoma in situ)
* Inability to consent
* Severe psychiatric illness
* Medical conditions impairing participation/adherence
* Non-adults, pregnant women, prisoners, and other legally protected vulnerable groups
* Dairy, soy, and/or fish allergy
* Non-English speaking
* Documented history of atrial fibrillation or other significant arrhythmias
* Receiving therapeutic anticoagulation (e.g., warfarin, direct oral anticoagulants) and/or clotting disorders (e.g., hemophilia, thrombocytopenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, approximately 18 months
  Calculated as the number of participants enrolled per month during the active recruitment period. Presented descriptively
Adherence Rate | From baseline (Week -2) to 3 months post-chemoradiotherapy
  The primary feasibility endpoint. Calculated as the proportion of enrolled participants who consume ≥75% of the prescribed supplement doses (2 bottles/day) throughout the intervention period, based on participant/caregiver tracking logs.
Retention Rate | From baseline (Week -2) to 3 months post-chemoradiotherapy
  Calculated as the proportion of enrolled participants who complete the intervention phase (through end of CRT) and the proportion who complete the 3-month post-CRT follow-up visit.
Adverse Events | From baseline (Week -2) to 3 months post-chemoradiotherapy
  Adverse event (AEs) means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Frequencies and percentages of all reported AEs will be tabulated by type, severity (CTCAE v5.0 grade), and investigator-assessed relatedness to the study supplement (Fresubin Supportan).
Supplement Acceptability | From baseline (Week -2) to 3 months post-chemoradiotherapy
  Assessed via structured questions during RDN visits and a final survey completed by the adult participant/caregiver.
Supplement Discontinuation due to AEs | From baseline (Week -2) through 3 months post-chemoradiotherapy
  The key safety endpoint. Calculated as the proportion of enrolled participants who discontinue the supplement due to an AE deemed at least possibly related to the supplement. A 95% binomial CI will be calculated for this proportion. The point estimate and CI will be compared to the pre-defined success threshold of <15%.

SECONDARY OUTCOMES:
Body composition | From baseline (Week -2) to 3 months post-chemoradiotherapy
  Skeletal Muscle Index as assessed using diagnostic CT images with sliceomatic software.
Nutrition Impact Symptoms | From baseline (Week -2) to 3 months post-chemoradiotherapy
  Change in patient-reported NIS will be assessed using the MDASI-HN total symptom severity score and relevant subscale scores.
Red Blood Cell Fatty Acid Profiles | From baseline (Week -2) to 3 months post-chemoradiotherapy
  Changes in key red blood cell (RBC) fatty acid levels (EPA, DHA, Arachidonic Acid, EPA:AA ratio)
FADS1/2 Genotyping | Baseline
  FADS1/2 Genotyping: Genotype frequencies (I/I, I/D, D/D for rs66698963) and allele frequencies (I allele, D allele) will be calculated and reported descriptively for the baseline samples. Exploratory analyses may examine outcomes stratified by genotype, but these will be hypothesis-generating only due to the small N.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen X, Beilman B, Gibbs HD, Hamilton JL, Parker N, Bur AM, Caudell JJ, Gan GN, Hamilton-Reeves JM, Jim HSL, Kirtane K, Lominska C, Crowder SL, Arthur AE. Nutrition in head and neck cancer care: a roadmap and call for research. Lancet Oncol. 2025 Jun;26(6):e300-e310. doi: 10.1016/S1470-2045(25)00087-7. PMID 40449504
- [Background] Morse RT, Ganju RG, Gan GN, Cao Y, Neupane P, Kakarala K, Shnayder Y, Lominska CE. Sarcopenia and Treatment Toxicity in Older Adults Undergoing Chemoradiation for Head and Neck Cancer: Identifying Factors to Predict Frailty. Cancers (Basel). 2022 Apr 22;14(9):2094. doi: 10.3390/cancers14092094. PMID 35565223
- [Background] Maino Vieytes CA, Mondul AM, Crowder SL, Zarins KR, Edwards CG, Davis EC, Wolf GT, Rozek LS, Arthur AE, On Behalf Of The University Of Michigan Head And Neck Spore Program. Pretreatment Adherence to a Priori-Defined Dietary Patterns Is Associated with Decreased Nutrition Impact Symptom Burden in Head and Neck Cancer Survivors. Nutrients. 2021 Sep 9;13(9):3149. doi: 10.3390/nu13093149. PMID 34579024
- [Background] Taha HM, Rozek LS, Chen X, Li Z, Zarins KR, Slade AN, Wolf GT, Arthur AE. Risk of Disease Recurrence and Mortality Varies by Type of Fat Consumed before Cancer Treatment in a Longitudinal Cohort of Head and Neck Squamous Cell Carcinoma Patients. J Nutr. 2022 May 5;152(5):1298-1305. doi: 10.1093/jn/nxac032. PMID 35170737
- [Background] Crowder SL, Douglas KG, Yanina Pepino M, Sarma KP, Arthur AE. Nutrition impact symptoms and associated outcomes in post-chemoradiotherapy head and neck cancer survivors: a systematic review. J Cancer Surviv. 2018 Aug;12(4):479-494. doi: 10.1007/s11764-018-0687-7. Epub 2018 Mar 20. PMID 29556926